CLINICAL TRIAL: NCT06795295
Title: Swallowing Dynamic of Two Implant Versus Single Implant Retained Mandibular Overdentures
Brief Title: Swallowing Dynamic of Implant Retained Mandibular Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Taha Abdo El_Baz, Clinical demonstrator, Prosthodontic Department, Faculty of dentistry, Mansoura University, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A05011122
Record Dates: First submitted 2025-01-20; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Swallowing
Keywords: swallowing dynamic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group І 2- IMOVD (Active Comparator): Patients received two implant on the mandibular canine regions to retain mandibular overdenture with locator attachment
  Interventions: Procedure: Implant retained mandibular overdenture
- Group ІІ 1-IMOVD (Active Comparator): Patients received single mandibular midline implant to retain mandibular overdenture with locator attachment
  Interventions: Procedure: Implant retained mandibular overdenture

INTERVENTIONS:
Procedure: Implant retained mandibular overdenture — Participants received dental implants to retain mandibular overdentures.
  Other Names: BTK implant

SUMMARY:
This Randomized clinical study was conducted to compare between two-implant versus single implant-retained mandibular overdenture regarding swallowing dynamic using The Test of Mastication and Swallowing Solids (TOMASS) and the Timed Water Swallow Test (TWST)

DETAILED DESCRIPTION:
There are lack of studies comparing single and two implant-retained mandibular overdentures regarding swallowing dynamic. This Randomized clinical study aimed to compare the effect of two treatment modalities of mandibular implant over denture on the swallowing dynamic.

8 completely edentulous patients were selected from the Out-Patient Clinic of Prosthodontics' Department, Faculty of Dentistry, Mansoura University seeking prosthetic rehabilitation. All patients were randomly distributed into two equal groups; Group I (Patients received two-implant mandibular overdenture with locator attachment) and Group II ( Patients received single implant mandibular overdenture with locator attachment) All subjects received a newly carefully constructed complete dentures and then the lower dentures were changed into mandibular implant retained overdentures using locator attachments by placing two implants on the mandibular canine regions for group I and single midline implant for group II.

Swallowing dynamic was evaluated after 3 months of complete denture insertion for both groups. After mandibular overdenture insertion swallowing dynamic was evaluated 2 weeks after insertion and three months after overdenture insertion for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Free from any systemic disease.
* Free from any medical or surgical conditions that cause dysphagia (swallowing problems).
* A sufficient residual alveolar bone quantity (height and width). This was verified by a CT scan using cone-beam computed tomography for each patient.
* All patients had sufficient bone either D2 or D3 by measuring the Hounsfield unit on CBCT scan.
* Residual ridges are covered by firm healthy mucosa.
* Class I maxilla-mandibular relationship.
* sufficient inter-arch space and restorative space for locator retained mandibular overdenture.

Exclusion Criteria:

* Patient with absolute contraindications for implant placement such as active cancer, immunosuppression, bleeding issues, and metabolic diseases that directly affect the bone such as osteoporosis, and hyperparathyroidism.
* Patients with relative contraindication: history of para functional habits such as bruxism, clenching, and bad habits such as smoking and alcoholism, uncontrolled diabetic patients.
* Patients with local contraindications for implant placement due to localized bone defects.
* Non-cooperative patients who don't follow instructions during and after the operation.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Swallowing Dynamic Of Two Implant Versus Single Implant Retained Mandibular Overdentures | The evaluation of swallowing by TOMASS for(no swallows, no of chews,and total time)was done after 3 months (3M-CD) of CD insertion, three months (3M-OD) after overdenture insertion.
  Evaluation of swallowing dynamic of both groups was done by The Test of Mastication and Swallowing Solids (TOMASS) to measure (number of swallows,number of chews,and total time)
Swallowing Dynamic Of Two Implant Versus Single Implant Retained Mandibular Overdentures | The evaluation of swallowing by TWST for (time per swallow, volume per swallow, and swallowing capcity) was done after 3 months (3M-CD) of CD insertion, three months (3M-OD) after overdenture insertion.
  swallowing dynamic of both groups was evaluated by the Timed Water Swallow Test (TWST) to measure (time per swallow, volume per swallow,and swallowing capcity)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura Universty, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No